CLINICAL TRIAL: NCT07193719
Title: Influence of Lung Volume Optimization Maneuver on Cardiac Output and Lung Mechanics in Children
Brief Title: Influence of Lung Volume Optimization Maneuver in Ventilated Children on Cardiac Output and Lung Compliance in Children With Congenital Heart Disease Undergoing Surgical Repair and on Prevention of Need for ECMO or Shortening of ECMO Duration in Children With Severe Respiratory Failure
Acronym: ILOCO
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Jan Clausen, Pediatric Cardiologist/Intensivist, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EA2/070/25
Record Dates: First submitted 2025-09-11; First posted 2025-09-26 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Congenital Heart Disease; Cardiopulmonary Bypass; Cardiac Surgery; Mechanical Ventilation; Positive End-expiratory Pressure (PEEP); Lung Volume; Lung Mechanics; Hemodynamic Changes; Children; ARDS; ECMO
Keywords: cardiopulmonary interactions; end-expiratory lung volume; PEEP titration
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: The type of intervention is one of clinical management (ventilatory management) and does not include a specific drug or biological
Who Masked: Outcomes Assessor
Masking Description: Statisticians
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Active Comparator): CHD study: This group receives so called standard of care. This includes relatively low levels of PEEP (5cmH2O in case of planned surgery) and no standardized PEEP titration
  ECMO study: This group receives so called standard of care. This includes PEEP of 10cmH2O, peak inspiratory pressures of 20cmH2O and no standardized PEEP titration
  Interventions: Procedure: Standard Care (in control arm)
- treatment (Experimental): CHD study: This group receives an individual lung volume optimization maneuver with PEEP titration. PEEP titration is performed while monitoring lung mechanics to optimize end-expiratory lung volume and find final "best PEEP".
  ECMO study: This group receives an individual lung volume optimization maneuver with PEEP titration during conventional or CDP titration with high frequency oscillatory ventilation. PEEP/CDP titration is performed while monitoring lung mechanics and EIT indices to optimize end-expiratory lung volume and find final "best PEEP/CDP".
  Interventions: Procedure: End-expiratory lung volume optimization maneuver with PEEP titration

INTERVENTIONS:
Procedure: End-expiratory lung volume optimization maneuver with PEEP titration — CHD study: PEEP titration (incremental/decremental) will be performed to optimize lung volume and find levels of PEEP corresponding to the best lung compliance at the end of surgery. Typically PEEP levels between 10-20cmH2O will be applied based on individual response of patients' lung mechanics. Tidal volume will be kept constant at 6ml/kg in cases and controls. Driving pressures will be limited to 15cmH2O. Balance of CO2 will be guaranteed by adjusting respiratory rate.
  ECMo study: PEEP/CDP titration (incremental/decremental) will be performed to optimize lung volume and find levels of PEEP/CDP corresponding to the best lung compliance, best match of overdistension and collapse and homogenization of tidal volume distribution (EIT) .
  Arms: treatment
Procedure: Standard Care (in control arm) — CHD study: Patients will receive pressure controlled ventilation with target tidal volume of 6ml/kg and PEEP of 5cmH2O. Driving pressures are limited to 15cmH2O. No LVOM will be applied.
  ECMO study: patients will receive standard ECMO ventilation (PEEP 10cmH2O and PiP 20cmH2O) without performing LVOM
  Arms: control

SUMMARY:
The goal of this randomized interventional clinical trial is to learn if a standardized lung volume optimization maneuver (LVOM) is beneficial in

1. study) children undergoing biventricular repair of their congenital heart disease (CHD) with cardiopulmonary bypass and
2. study) in children with severe respiratory failure at risk for or need for ECMO.

The main questions it aims to answer are:

Main hypotheses of CHD study: Does a standardized PEEP-Titration maneuver, to optimize end-expiratory lung volume improve:

* cardiac performance
* lung function

Does it make a difference in:

* length of ventilation
* ventilation/perfusion mismatch of the lung
* need for vasopressor support?

Main hypotheses of ECMO study:

Does a LVOM in children/infants with severe respiratory failure /ARDS

* improve lung compliance and gas exchange
* facilitate lung protective ventilation according to PALICC-2 guidelines
* improve lung aeration and V/Q-matching assessed with EIT

Does it make a difference in

* need for ECMO
* duration of ECMO runs
* hemodynamics stability

DETAILED DESCRIPTION:
1) The objective of the CHD study is to define the impact of a LVOM after cardiac surgery with CPB on hemodynamics and lung mechanics in children with congenital heart disease (CHD) undergoing surgery.

The Specific Aims of this work are:

Specific Aim 1:

Evaluate hemodynamics and lung mechanics during and after a LVOM:

In cases of children undergoing cardiac surgery all measurements will be performed with closed chest conditions.

Specific Aim 2:

Evaluate a potential benefit of lung volume optimization by performing PEEP titration on hemodynamics and lung mechanics compared to standard care without PEEP titration to optimize end-expiratory lung volume while maintaining same tidal volume targets in cases and controls.

Hypotheses:

1. Hemodynamics and lung mechanics will be significantly different before and after LVOM. We expect that there will be little difference between intervention and control group before performing PEEP titration in the interventional group.
2. Once the PEEP titration has been performed in the interventional group, we hypothesize that patients who received the intervention will have improved hemodynamics and lung mechanics with modest PEEP while receiving the same tidal volume than the control group (U-shaped curves).

Rationale: Surgery with cardiopulmonary bypass typically involves an interruption of mechanical ventilation while CPB is running. This is oftentimes associated with atelectasis formation and impaired gas exchange due to reduced end-expiratory lung volume. While there have been few studies in adults that have shown that optimization of lung volume by performing PEEP titration after CPB can significantly improve Cardiac Index and right ventricular function, there have been only very few prospective pediatric studies which assessed the impact of different PEEP settings on hemodynamics, and lung mechanics after cardiac surgery in children. Because these patients are generally among the most fragile postoperative patients, it is critical to understand if specific ventilator strategies can help mitigate any negative hemodynamic consequences after surgery. The purpose of this study is to understand the critical cardiopulmonary interactions that occur with changes in lung volumes, and to determine optimal approaches to mechanical ventilation under these different circumstances.

Cardiopulmonary interactions differ based on the underlying cardiac anatomy and physiology. Most studies of cardiopulmonary interactions following surgery for congenital heart disease have examined the difference between positive and negative pressure ventilation. This work consistently showed improvement in cardiac output and pulmonary blood flow with negative pressure ventilation, while positive pressure ventilation was associated with decreased cardiac output. However, these studies have been conducted in the 1990's and positive pressure ventilation has changed significantly in the meantime.

Similarly, while patients with left ventricular dysfunction generally benefit from positive pressure ventilation, there is little data regarding the hemodynamic effects of positive pressure ventilation on right ventricular performance.

Modulating pulmonary vascular resistance by optimizing lung volumes might be a promising approach to improve both lung mechanics and hemodynamics. Studies in this population have focused more on the effects of FiO2 and hyperventilation than on respiratory mechanics and cardiopulmonary interactions.

2) The objective of the ECMO study is to evaluate if a LVOM in children and infants with ARDS at risk or need for ECMO has an impact on ECMO prevention or shortening of ECMO duration.

Specific aims:

* assess the effect of LVOM on lung aeration and perfusion assessed with EIT
* assess the effect of LVOM on hemodynamics with (primarily VV-ECMO) and without ECMO
* evaluate if LVOM can prevent the need for ECMO
* evaluate if LVOM can shorten ECMO duration

Rationale:

Children with NARDS or PARDS usually have reduced lung volumes. Typically ECMO is initiated when oxygenation index approaches 40 with further deterioration of hypercarbia, hemodynamics and worsening hypoxemia. Current treatment strategies include reducing ventilatory support on ECMO ("rest settings") which is typically followed by a "whiteout" of the lungs reflecting lung collapse and fluid infiltration. Usually within 10 days of ECMO support invasive ventilation is gradually increased to re-open the lung and allow for ECMO weaning. Optimizing lung volumes by performing a LVOM early on in the disease process might be beneficial to wean ECMO faster or even prevent its need by avoiding massive lung collapse during rest settings in patients that have high potential for lung recruitability.

ELIGIBILITY:
CHD study:

Inclusion Criteria

* congenital heart disease
* surgery with cardiopulmonary bypass

Exclusion Criteria:

* single ventricle physiology
* ECMO/VAD
* <36weeks of gestational age
* chronic lung disease
* Endotracheal tube leak > 15%
* lack of informed consent from parents.

ECMO study Inclusion Criteria

* patients with respiratory failure on ECMO or at risk for ECMO
* invasive ventilation

Exclusion Criteria:

- severe lung hypoplasia or interstitial lung disease

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-12-05 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-12-20 (Estimated)

PRIMARY OUTCOMES:
CHD study: Cardiac Index (L/min/BSA) 2. ECMO study: shortening of ECMO duration (Hours) | perioperatively/periprocedurally
  CHD study: assessed by using POCUS ECMO study: time course (Hours)

SECONDARY OUTCOMES:
lung mechanics | perioperatively/periprocedurally
  lung compliance (ml/cmH2O/kg)
right ventricular performance | perioperatively/periprocedurally
  TAPSE PAAT Strain
Ventilation distribution | perioperatively/periprocedurally
  EIT
Lung perfusion | perioperatively/periprocedurally
  assessed with EIT (electrical impedance tomography)
dead space | perioperatively/periprocedurally
  pulmonary dead-space fraction (Vd/Vt)
avDO2 | perioperatively/periprocedurally
  difference in arteriovenous oxygen content

CONTACTS AND LOCATIONS:
Locations (1):
- German Heart Center of the Charité, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided